CLINICAL TRIAL: NCT04779788
Title: I-125 Seeds Loaded Stent Insertion for Inoperable Hilar Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210218015
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Hilar Cholangiocarcinoma
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-125 seeds loaded stent group (Experimental): Patients who receive the I-125 seeds loaded stent insertion
  Interventions: Device: I-125 seeds loaded stent (self-expanded metal stent with I-125 seeds, Micro-Tech, Nanjing, China)
- Normal stent group (Active Comparator): Patients who receive the normal stent insertion
  Interventions: Device: Normal stent (self-expanded metal stent without I-125 seeds, Micro-Tech, Nanjing, China)

INTERVENTIONS:
Device: I-125 seeds loaded stent (self-expanded metal stent with I-125 seeds, Micro-Tech, Nanjing, China) — An I-125 seeds loaded stent consisted of two overlapped parts: an inner normal bare stent and an outer seeds-loaded stent
  Arms: I-125 seeds loaded stent group
Device: Normal stent (self-expanded metal stent without I-125 seeds, Micro-Tech, Nanjing, China) — Bare self-expanded metal stent
  Arms: Normal stent group

SUMMARY:
Malignant biliary obstruction usually arise in patients suffering from primary or metastatic hepatobiliary tumors. Approximately 80% of malignant biliary obstruction patients are not eligible for surgical resection, and as such palliative stent insertion is the only treatment option available for most patients. At present, I-125 seeds loaded stent has been developed to improve the stent patency and patients' survival. Hilar malignant biliary obstruction is an important part of malignant biliary obstruction. Hilar cholangiocarcinoma is the most common disease which causes hilar malignant biliary obstruction. Herein, we assessed the clinical and long-term efficacy of I-125 seeds loaded stent insertion for hilar cholangiocarcinoma patients.

DETAILED DESCRIPTION:
Malignant biliary obstruction usually arise in patients suffering from primary or metastatic hepatobiliary tumors. Approximately 80% of malignant biliary obstruction patients are not eligible for surgical resection, and as such palliative interventions are the only treatment option available for most patients. Of the available palliative treatments, percutaneous or endoscopic stent insertion is the most frequently used to treat malignant biliary obstruction patients.

Although stent insertion can achieve the good short-term outcomes for patients with malignant biliary obstruction, stent dysfunction remains a common outcome in these treated patients, limiting the long-term efficacy of this treatment strategy. In order to overcome this shortcoming of the normal stent insertion, many researchers have developed a novel biliary I-125 seeds loaded stent. The I-125 seeds loaded stents not only can effectively relieve the jaundice, but also can provide the brachytherapy to the tumor. Previous meta-analyses also indicated that showed that relative to normal stent insertion, I-125 seeds loaded stent insertion was associated with longer survival and stent patency in inoperable malignant biliary obstruction patients. However, most previous studies included malignant biliary obstruction patients with different cancer types and malignant biliary obstruction sites, and therefore, the risk of bias did exist. Therefore, there is a clear need for a study comparing these two stent types in patients with a single type of cancer.

Hilar malignant biliary obstruction is an important part of malignant biliary obstruction. Hilar cholangiocarcinoma is the most common disease which causes hilar malignant biliary obstruction. Herein, we assessed the clinical and long-term efficacy of I-125 seeds loaded stent insertion for hilar cholangiocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosed hilar Cholangiocarcinoma; Inoperable cases; Patients showed evidence of obstructive jaundice; Eastern Cooperative Oncology Group performance status < 4.

Exclusion Criteria:

Patients who underwent post-operative external radiotherapy; Patients in whom prior biliary stent insertion or drainage were performed; Patients suffering from serious dysfunction of the pulmonary, renal, cardiac, or coagulatory systems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization until the date of first documented death from any cause, assessed up to 12 months
  From the date of randomization until the date of first documented death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Chi Li, MD, Principal Investigator — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Chen G, Zhang M, Sheng YG, Yang F, Li ZQ, Liu TG, Fu YF. Stent with radioactive seeds strand insertion for malignant hilar biliary obstruction. Minim Invasive Ther Allied Technol. 2021 Dec;30(6):356-362. doi: 10.1080/13645706.2020.1735446. Epub 2020 Mar 3. PMID 32125207
- [Background] Yang S, Liu Y, Teng F, Wu AL, Lin J, Xian YT, Xu YS. Radioactive Stent Insertion for Inoperable Malignant Common Biliary Obstruction. Surg Laparosc Endosc Percutan Tech. 2020 Aug 5;31(1):61-65. doi: 10.1097/SLE.0000000000000848. PMID 32769739